CLINICAL TRIAL: NCT02111161
Title: Immunoglobulin for Necrotizing Soft Tissue Infections: a Randomised Controlled Trial
Acronym: INSTINCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Anders Perner (Other)
Collaborators: CSL Behring (Industry)
Responsible Party: Sponsor-Investigator, Anders Perner, MD, PhD, Professor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RH4131-03
Record Dates: First submitted 2014-04-03; First posted 2014-04-11 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Necrotizing Soft Tissue Infection; Necrotizing Fasciitis; Gas Gangrene; Fournier Gangrene
Keywords: Randomised controlled trial (RCT); Immunoglobulin; Patient Reported Outcome; Health-Related Quality of Life; Short Form-36 (SF-36)
MeSH Terms: conditions — Fasciitis, Necrotizing; Gas Gangrene; Fournier Gangrene | interventions — Immunoglobulins, Intravenous; Immunoglobulin G; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IVIG (Privigen) (Active Comparator): Intravenous polyspecific immunoglobulin G (Privigen). Dosage: 25 g/day (250 ml) for three consecutive days
  Interventions: Drug: IVIG (Privigen)
- Saline 0.9% (Placebo Comparator): 0.9% saline for Intravenous administration. Dosage: 250 ml for three consecutive days.
  Interventions: Drug: Saline 0.9%

INTERVENTIONS:
Drug: IVIG (Privigen) — Three doses of 25 g IVIG (250 ml)
  Other Names: Privigen; Immunoglobulin G
  Arms: IVIG (Privigen)
Drug: Saline 0.9% — Three doses of Saline 0.9% (250 ml)
  Other Names: NaCl
  Arms: Saline 0.9%

SUMMARY:
The purpose of this study is to estimate the effect of intravenous polyspecific immunoglobulin G (IVIG) compared with placebo (saline) on the patient-reported outcome measure Physical Component Summary Score (PCS) of the SF-36 in patients with necrotizing soft tissue infections (NSTI).

DETAILED DESCRIPTION:
Patients with necrotizing soft tissue infections (NSTI) receive intravenous polyspecific immunoglobulin G (IVIG) as part of the standard treatment at Rigshospitalet. The current evidence available does not support neither the use of IVIG, nor omitting it, as adjuvant treatment of NSTI. With this trial the investigators will estimate the effects of IVIG on a patient-reported outcome and other important outcomes in patients with NSTI

Design A randomized, double-blinded, clinical trial where patients are randomly assigned 1:1 to receive either IVIG or an equal volume of 0.9% saline.

Location A single centre trial conducted at Dept. of Intensive Care 4131, Copenhagen University Hospital, Rigshospitalet.

Randomisation Randomisation will be stratified according to primary presentation of NSTI on the extremities/head/neck (yes/no) as streptococci mainly affect these anatomical sites. Two randomisation lists, with varying block size, are generated. Two separate boxes contain sequentially numbered, opaque, sealed envelopes (SNOSE). Two people independent of the trial will generate the envelopes following the randomisation lists and will document that the envelopes are concordant with the randomisation lists. Staff at trial site will have access to the boxes around the clock, and will draw an envelope containing a patient randomisation- and medicine log document assigned either "Privigen" or "Saline" from one of the two boxes.

Intervention Trial medicine is given when the patient arrives at the ICU and the following two consecutive days. Alternatively, the first dose of trial medicine will be given in the operating theatre.The trial medicine will consist of either IVIG 25 g/day (250 ml) (Privigen, CSL Behring) or an equal volume of 0.9% saline. The dosage of IVIG is 25g/day for three consecutive days for all patients, which is according to the clinical protocol at Rigshospitalet. The treatment will be given according to the clinical protocol for Privigen at Rigshospitalet. The treating clinicians will decide all other interventions.

Blinding The trial medicine will be prepared in the ICU at the time of arrival of the patient and the following two consecutive days by an ICU nurse not otherwise involved in the care of the trial patient and is supervised by another staff member who as well is not involved in the care of the patient. Privigen has a slight yellowish appearance whereas saline is clear. Furthermore, Privigen is produced in bottles of 50 and 100 ml, respectively. A bottle of Privigen will be packed with a bag of saline, containing a corresponding number of millilitres, in a black plastic bag and sealed with a plastic strip. An orange, transparent infusion set (B. Braun, ref. 8700127SP) is inserted into either the Privigen bottle or the bag containing saline, dependent on whether the patient has been allocated to active treatment or placebo. The orange colour masks the fluid colour while allowing air bubbles to be seen. A piece of non-transparent tape will mask the drip chamber making it impossible to see the frothing of Privigen. For each of the three dosages of trial medicine, three bags are prepared, containing 100 ml, 100 ml and 50 ml respectively. The bag will be marked with an etiquette containing the patient number. If unblinding is necessary, this is easily done by looking in the envelope with the same patient number.

Medicine score The trial medicine batch number will be noted on the patient randomisation- and medicine log document by the ICU nurse preparing the trial medicine. The attending physician will prescribe "trial medicine" in the electronic medication file (CIS 3.9.1, Daintel).

Subgroup Analysis Presumed Streptococcal Infection A subgroup analysis will be performed on patients with primary presentation of NSTI on the extremities, neck or head as these are more likely to be streptococcal infections, in which the effects of IVIG may be different.

Data Registration Data will be entered into the electronically, web-based case report form (eCRF) from patient notes by trial personnel. The eCRF is specifically designed for this purpose.

Safety

Patients will be withdrawn from the trial protocol if the following occurs:

* SARs or SUSARs Patients withdrawn from the trial for the above mentioned reasons will receive the standard protocol treatment for NSTI with the exception of IVIG.

During the trial, Sponsor will send yearly reports on the occurrence of SARs to the Danish Health and Medicines Authority and Regional Ethics Committee.

Suspected Unexpected Serious Adverse Reactions Suspected unexpected serious adverse reactions (SUSARs) will be defined as serious adverse reactions not described in the summary of product characteristics (SPC) for Privigen (no serious adverse reactions are described for 0.9% saline). Sponsor will report any SUSARs within 7 days to the Danish Health and Medicines Authority via Eudravigilance Clinical Trials Module, to the Regional Ethics Committee and to CSL Behring. During the trial, investigator will send yearly reports on the occurrence of SUSARs to the Danish Health and Medicines Authority and the Regional Ethics Committees.

Adverse Events and Serious Adverse Events Adverse events (AEs) and serious adverse events (SAEs) will not be recorded as an entity because the majority of ICU patients will experience several SAEs during their critical illness. In addition, most SAEs will be captured in the secondary outcome measures (SOFA scores and bleeding).

Termination of Trial The trial will be terminated prematurely in the case that new, definite information regarding the use of IVIG in patients with NSTI arises.

Sample Size Estimation 50 subjects in each group are needed to detect a difference of 7 points in PCS of SF-36 based on an expected score of 42 (SD 11) in the control group (data from our own follow-up studies), for a power of 80% and a two-tailed significance level of 0.05, and an expected 1-year mortality rate of 20%.

Statistical Methods Analysis will be by intention-to-treat comparing PCS of SF-36 in the two groups after six months by chi-squared test and multiple logistic regression analysis using unadjusted analyses and analyses adjusted for patient variables (SAPS II and SOFA score in the 24 h prior to randomisation).

Patients Included In Final Statistical Analysis Patients who are withdrawn from the trial protocol will be followed up and analysed as the remaining patients. Patients who are transferred to another ICU will be followed up for the primary outcome measure. Patients who are withdrawn will not be replaced by new patients, with the exception of the specific case, where the patient demands deletion of all registered data.

Accountability Procedure for Missing Data Imputation will be used if missingness >5%.

Interim Analysis An interim analysis will not be performed as analyses of a sample size below the planned 100 patients are less meaningful for those outcomes that are of relevance (mortality and SARs).

Monitoring

We will perform Good Clinical Practice (GCP)-monitoring according to a predefined monitoring plan including the following issues:

* Initiation visit
* For all patients: Documented informed consent
* Inclusion and exclusion criteria
* Documented delivery or non-delivery in the eCRF of the intervention according to the protocol compared with source data being patients' hospital records
* Termination visit: Primary outcome

Data Handling and Record Keeping Data will be handled according to the National Data Protection Agency, and is protected by the national law "Loven om behandling af personoplysninger" and "Sundhedsloven". All original records (incl. consent forms, eCRFs, and relevant correspondences) will be archived at trial site for 15 years. The clean electronic trial database file will be delivered to the Danish Data Archive and maintained for 15 years and anonymised if requested by the authorities.

Quality Control and Quality Assurance The subinvestigator will be responsible for preparing the research nurses and other trial site personnel before the initiation of the trial. This education will be continuously documented.

Monitoring of the Intervention Groups Day-to-day monitoring of the eCRF will be done by persons delegated to this specific task.

Ethics The trial will adhere to the Helsinki Declaration and Danish law. Inclusion will start after approval by the Regional Ethics Committee, the Danish Health and Medicines Authority and the National Data Protection Agency (via the Joint Notification System of The Capital Region of Denmark - Region Hovedstaden) and trial registration at www.clinicaltrials.gov.

ELIGIBILITY:
Inclusion Criteria:

* Necrotizing soft tissue infection (NSTI) based on surgical findings
* Age >18 years
* Admitted to or planned to be admitted to the ICU at Rigshospitalet (RH)

Exclusion Criteria:

* >48 hour from the primary diagnosis to arrival at RH
* More than one dose of IVIG given within current admission
* Known hypersensitivity to IVIG
* Hyperprolinaemia (obtained from hospital notes)
* Pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-04; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Physical Component Summary Score (PCS) of Short-Form 36 (SF-36) | Six months after randomisation

SECONDARY OUTCOMES:
Mortality | 28, 90 and 180 days
Time to resolution of shock | During ICU admission (expected average of 8 days)
  Maintenance of a systolic blood pressure of at least 90 mmHg without vasopressor support for 24 hours
Severe bleeding | During ICU admission (expected average of 8 days)
  Clinical bleeding and use of 3 units of red blood cells (RBCs) within 24 hours at any time in the ICU
Any bleeding in the ICU | During ICU admission (expected average of 8 days)
Use of blood products | During ICU admission
  Total volumes during the ICU admission
SOFA scores (AUC), excluding the Glasgow Coma Score (GCS) score | Day 1-7
Use of renal replcement therapy (RRT), ventilation and vasopressor in the ICU | During ICU admission (expected average of 8 days)
Days alive off life support in the 90 days after randomisation | 90 days after randomisation
Days alive and out of hospital in the 180 day follow-up period | 180 day follow-up period
Amputation, any location | Within 180 days
Serious Adverse Reactions (SARs) in the ICU | During ICU admission (expected average of 8 days)
  * Allergic reactions
  * Haemolytic anaemia
  * Aseptic meningitis syndrome
  * Thrombus
  * Transmittable agents
  * Acute kidney injury

CONTACTS AND LOCATIONS:
Overall Officials: Anders Perner, Professor, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Dept. of Intensive Care 4131, Copenhagen University Hospital, Rigshospitalet, Copenhagen, Danmark, Denmark

REFERENCES:
- [Derived] Bergsten H, Madsen MB, Bergey F, Hyldegaard O, Skrede S, Arnell P, Oppegaard O, Itzek A, Perner A, Svensson M, Norrby-Teglund A; INFECT Study Group. Correlation Between Immunoglobulin Dose Administered and Plasma Neutralization of Streptococcal Superantigens in Patients With Necrotizing Soft Tissue Infections. Clin Infect Dis. 2020 Oct 23;71(7):1772-1775. doi: 10.1093/cid/ciaa022. PMID 31916575
- [Derived] Madsen MB, Hjortrup PB, Hansen MB, Lange T, Norrby-Teglund A, Hyldegaard O, Perner A. Immunoglobulin G for patients with necrotising soft tissue infection (INSTINCT): a randomised, blinded, placebo-controlled trial. Intensive Care Med. 2017 Nov;43(11):1585-1593. doi: 10.1007/s00134-017-4786-0. Epub 2017 Apr 18. PMID 28421246
- [Derived] Madsen MB, Lange T, Hjortrup PB, Perner A. Immunoglobulin for necrotising soft tissue infections (INSTINCT): protocol for a randomised trial. Dan Med J. 2016 Jul;63(7):A5250. PMID 27399982